CLINICAL TRIAL: NCT05860556
Title: Sustainable Eating Pattern to Limit Malnutrition in Older Adults (SENIOR)
Brief Title: Sustainable Eating Pattern to Limit Malnutrition in Older Adults
Acronym: SENIOR
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pavia (Other)
Collaborators: Fondazione Salvatore Maugeri (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Hellas Cena, Pro-Rector for Third Mission; Professor of Dietetics and Clinical Nutrition; Human Nutrition Researcher and Head of the Clinical Nutrition Laboratory, University of Pavia
Other Study IDs: 21042023; CUP: F13C22001210007 (Other Grant/Funding Number: PNRR - MUR)
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Malnutrition; Sarcopenia
Keywords: GLIM; older adults; prevalence; hospital; nutrition; risk factor; malnutrition; sarcopenia; sustainability
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SENIOR STUDY is aimed at improving the condition of older adults and malnutrition management in and out Italian hospital settings, since malnutrition is highly prevalent, clinically relevant and potentially treatable condition. This study consist of two phases: an initial cross-sectional phase and a secondary nutritional intervention phase (RCT).

The SENIOR CROSS-SECTIONAL study aims to map malnutrition status in accordance with the most recent GLIM criteria and investigate the association between malnutrition and anthropometric, demographic and socioeconomic, and lifestyle factors. In addition, sarcopenia will be diagnosed (EWGSOP2 consensus criteria) and blood markers will be measured.

Malnutrition in Italian hospital setting is highly prevalent but the current malnutrition data prevalence and the general characteristics of older adults are not updated. Thus, it is expected to find a high malnutrition prevalence and an inadequate nutritional status.

DETAILED DESCRIPTION:
The SENIOR cross-sectional study is a multicenter study conducted in two North Italian Scientific Hospitalization and Treatment Institution in Pavia on older adults (≥ 65 years old). The estimated duration is 36 months with an preferred starting date on September 2023.

The primary objective of the SENIOR cross-sectional is the evaluation of the nutritional status in at least a total of 200 free-living and hospitalized older adults. Therefore, the primary endpoint is to define the malnutrition prevalence in free-living and hospitalized older adults with GLIM criteria, which is the most update recent international consent.

As secondary objectives, a mapping of other relevant factors potentially associated with malnutrition will be carried out on the population target: lifestyle, socioeconomic status, anthropometric measures, clinical condition including medical treatment and blood analysis. In addition, the impact of these factors on health status of the target population will be investigated, potentially leading to the identification of new malnutrition risk factors.

To the over 65 older adults, admitted at the two hospitals for medical visits or recovery, will be proposed to participate to the SENIOR cross-sectional study. After the participants' signature of the informed consent, the clinical and pathological information will be gathered to assess the eligibility.

On eligible subject different variables will be measured. Dietary habits will be evaluated through a Mediterranean diet questionnaire (MEDI-LITE) and the MIND diet questionnaire. Physical activity will be evaluated with the Physical Activity Scale for the Elderly (PASE) questionnaire and, if the subject has physical limitation, with the Barthel Index. Sleep quality will be investigated with Pittsburgh questionnaire. Emotional status of participants will be examined with the Geriatric Depression Scale 15 item (GDS-15). Quality of life will be measured with SF-12 questionnaire.

Anthropometric variables include weight, height (knee height and demi-span), waist circumference, and body composition (bioimpedance analysis, BIA). In addition, strength (handgrip) and locomotion (gait speed) will be evaluated. Strength (handgrip), Appendicular Skeletal Mass (ASM) and locomotion (gait speed) are necessary to diagnose sarcopenia according to the European Working Group on Sarcopenia in Older People 2 (EWGSOP2) consensus. Intrinsic capacity is a score developed by the World Health Organisation (WHO) which capture the psychological and physical condition of the older adults. In this study four out of five dimensions of the intrinsic capacity will be evaluated: locomotion, vitality, cognition and psychological.

Blood analysis will be carried out on a subgroup to evaluate the participants' inflammatory, nutritional and clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Admission to U.O. of General Medicine and to U.O.S.D. of Endocrinology and Metabolic diseases of two Scientific Hospitalization and Treatment Institutions of Pavia, Italy
* Informed consent written and signed

Exclusion Criteria:

* Dysphagia
* Prior nutritional medical treatment
* Terminal disease
* History of gastric bypass, anorexia nervosa, liver failure
* Dementia or severe confusion (MMSE score <24/30)
* Patients with tumor diagnosis not in remission and currently not treated with oncological therapy
* Patients with chronic or acute respiratory failure

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults (over 65 years old), free-living or hospitalized, admitted at the hospitals
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of malnutrition in free-living and hospitalized older adults | Day 1
  Malnutrition diagnosis (GLIM) with Malnutrition Universal Screening Tool (MUST) screening tool

SECONDARY OUTCOMES:
Prevalence of sarcopenia in free-living and hospitalized older adults | Day 1
  Sarcopenia diagnosis (EWGSOP2)
Level of physical activity in free-living and hospitalized older adults | Day 1
  Physical Activity Scale for the Elderly questionnaire. Total score ranges from 0 to 450 and an higher score represents a higher level of physical activity.
  OR Barthel Index. The total score ranges from 0 to 100. The lower score indicates a totally dependent and a higher score indicates a higher independence in daily activities
Level of adherence to Mediterranean diet in free-living and hospitalized older adults | Day 1
  Medi-Lite adherence score questionnaire. Total score ranges between 0-18. A high score represents a higher adherence to Mediterranean diet
Level of adherence to Mind Diet in free-living and hospitalized older adults | Day 1
  Mind diet score. Total score ranges from 0 to 15. A higher score indicate a higher adherence to Mind Diet
Sleep quality in free-living and hospitalized older adults | Day 1
  pittsburgh sleep quality index. Total score ranges between 0-21. A higher score represents higher sleep difficulties
Level of quality of life in free-living and hospitalized older adults | Day 1
  Short-Form Health Survey 12. Total score ranges between 0-100. A higher score represents a better quality of life
Level of depression in free-living and hospitalized older adults | Day 1
  Geriatric Depression Scale. Total score ranges between 0-15. A higher score represents higher depression status
Level of intrinsic capacity in free-living and hospitalized older adults | Day 1
  * Locomotion (4 m gait speed) (m/s); score ranges between 0-2
  * Vitality (malnutrition according to GLIM criteria); score ranges between 0-2
  * Cognition (Mini Mental State Examination); score ranges between 0-2
  * Psychological state (geriatric depression scale); score ranges between 0-2 The scores of the precedent domains will be summarized to calculate the intrinsic capacity total score, which ranges from 0 to 8. A higher score represents a higher intrinsic capacity
Potential correlation between blood biomarkers and malnutrition in free-living and hospitalized older adults | Day 1
  Biomarkers blood measured from fasting blood samples are:
  Complete blood count with leukocyte count Lipid profile (Low density lipoprotein, high density lipoprotein, total cholesterol, triglycerides) (mg/dl) C reactive Protein (CRP) (mg/dl) Plasmatic creatinine (mg/dl) Transaminases (glutamic oxaloacetic transaminase, Glutamic-Pyruvic Transaminase, gamma-glutamyl transferase) (U/I) Alkaline phosphatase (U/L) Creatin Kinase (UI/L) Prealbumin (g/mL) Cytokine (interleukin-1β, interleukin-6, interleukin-10, tumor necrosis factor-α, transforming tumor factor-β) Glycemia (mg/dl) Insulin (µU/mL) Homocysteine (µmol/L) Vitamines (D, B12, B9) Minerals (Na, K, Mg, Ca, Fe, Zn)
Socio-demographic characteristic in free-living and hospitalized older adults | Day 1
  Structured interview (sex, age, ethnicity, level of education, socioeconomic status, number of people in the house, type of job)

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, Prof, Principal Investigator — Laboratory of Dietetics and Clinical Nutrition, Department of Public Health, Experimental and Forensic Medicine, University of Pavia; Clinical Nutrition and Dietetics Service, Unit of Internal Medicine and Endocrinology, Pavia; Flavia Magri, Prof, Principal Investigator — Department of Internal Medicine and Therapeutics, University of Pavia and Istituti Clinici Scientifici Maugeri IRCCS, Unit of Internal Medicine and Endocrinology; Istituti Clinici Scientifici Maugeri IRCCS, Unit of Endocrinology and Metabolism; Antonio Di Sabatino, Prof, Principal Investigator — Department of Internal Medicine and Therapeutics, University of Pavia; Fondazione IRCCS Policlinico San Matteo, Internal Medicine Unit, Pavia